CLINICAL TRIAL: NCT06994650
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of HRS9531 Injection in Subjects With Obstructive Sleep Apnea (OSA) and Obesity Who Are on Positive Airway Pressure Ventilation (PAP) Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS9531-307
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-05

CONDITIONS: Subjects With Moderate-to-severe OSA and Obesity Who Are on PAP Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS9531 (Experimental)
  Interventions: Drug: HRS9531
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS9531 — HRS9531 will be administered by Subcutaneous injection
  Arms: HRS9531
Drug: Placebo — Matching Placebo will be administered by Subcutaneous injection
  Arms: Placebo

SUMMARY:
This study is a phase 3 clinical trial, aiming to evaluate the efficacy and safety of HRS-9531 injection in obese subjects with obstructive sleep apnea (OSA) who are on positive airway pressure ventilation (PAP) therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 -75 (inclusive), male or female Sex
2. BMI ≥28.0 kg/m2；
3. ≥3 months of diet/exercise control pre-screening with ≤5.0 kg weight fluctuation in prior 3 months.
4. Confirmed OSA diagnosis with screening PSG showing AHI ≥15.0 events/h.
5. ≥3 months of PAP therapy pre-screening with planned continuation; willingness to pause PAP ≥1 week before each PSG.
6. Females/males of childbearing potential must use highly effective contraception from consent until 2 months post-treatment, with no pregnancy/donation plans. Females require negative pregnancy test ≤3 days pre-randomization and non-lactating.

Exclusion Criteria:

1. Endocrine disorders significantly affecting weight (e.g., Cushing's syndrome, hypo-/hyperthyroidism) or monogenic/hereditary obesity syndromes excluded.
2. Diabetes mellitus (excluding gestational diabetes).
3. Prior/planned OSA-related major surgeries (e.g., tonsillectomy/adenoidectomy) that may affect breathing.
4. Have significant craniofacial abnormalities that may affect breathing at baseline
5. Have diagnosis of Central or Mixed Sleep Apnea with % of mixed or central apneas/hypopneas ≥50%, or diagnosis of Cheyne Stokes Respiration
6. Respiratory and neuromuscular diseases that could interfere with the results of the trial in the opinion of the investigator.
7. Impaired gastric emptying (e.g., gastric bypass, pyloric stenosis)；Chronic use of GI motility-affecting drugs；Severe GI disorders (e.g., active PUD, IBD)；GI surgeries (except non-motility-affecting procedures)
8. Pancreatic disorders (acute/chronic pancreatitis, pancreatic injury)；Acute cholecystitis history；Symptomatic/treated gallbladder disease
9. Have used drugs or treatments that may cause significant weight gain or loss within 3 months
10. Investigator-determined unsuitability/unwillingness to pause PAP therapy for at least 1 week pre-PSG (e.g., safety/occupational/personal considerations).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The change of AHI form baseline after 52 weeks of treatment | 52 weeks

SECONDARY OUTCOMES:
The percentage change in AHI from baseline after 52 weeks of treatment | 52 weeks
The percentage of subjects with ≥50% AHI reduction from baseline after 52 weeks of treatment; | 52 weeks
The percentage of subjects with AHI <5.0 events /h, or AHI ranging from 5.0 to 14.0 events/h and Epworth Sleepiness Scale (ESS) ≤10 after 52 weeks of treatment; | 52 weeks
The percent change in body weight from baseline after 52 weeks of treatment. | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided